CLINICAL TRIAL: NCT06055673
Title: Angiotensin Converting Enzyme rs (1799752) Gene Polymorphism and Development of In-Stent Restenosis in Patients With Stable Coronary Artery Diseases in Sohag Hospital University.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud Kadry, lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-09-9PD
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Angiotensin Converting Enzyme rs (1799752) Gene Polymorphism and Development of In-Stent Restenosis in Patients With Stable Coronary Artery Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA EXTRACTION
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: patients with ISR confirmed by coronary angiography
  Interventions: Genetic: DNA extraction AND Real- time polymerase chain reaction analysis to POLYMORPHISM OF in in-stent restenosis (ISR) in CAD
- patients without restenosis non ISR group
  Interventions: Genetic: DNA extraction AND Real- time polymerase chain reaction analysis to POLYMORPHISM OF in in-stent restenosis (ISR) in CAD

INTERVENTIONS:
Genetic: DNA extraction AND Real- time polymerase chain reaction analysis to POLYMORPHISM OF in in-stent restenosis (ISR) in CAD — Real- time polymerase chain reaction a gene polymorphism in in-stent restenosis (ISR) in CAD.
  Other Names: genotyping of angiotensin converting enzyme in in-stent restenosis

SUMMARY:
One of the most common medical approaches to the treatment of coronary artery disease (CAD) is the percutaneous coronary intervention (PCI) which became frequent due to high efﬁciency and safety of this procedure. Modern-day advances in pharmacotherapy and the device innovations over the last thirty years enhanced the benign outcomes of patients with unstable or multivessel CAD, and multiple co-morbidities, treated by PCI .

In-stent restenosis (ISR) is a recognized complication following percutaneous coronary intervention in which the luminal diameter is narrowed through neointimal hyperplasia and vessel remodeling. Although rates of ISR have decreased in most recent years owing to newer generation drug-eluting stents, thinner struts, and better intravascular imaging modalities, ISR remains a prevalent dilemma that proves to be challenging to manage. Several factors have been proposed to contribute to ISR formation, including mechanical stent characteristics, technical factors during the coronary intervention, and biological aspects of drug-eluting stents .identiﬁcation of risk factors and mechanisms underlying ISR is necessary for understanding the process, the risk stratiﬁcation, and optimal treatment development. Restenosis, as a physiological response to mechanical damage, involves two mechanisms which are neointimal hyperplasia and vessel remodeling [3]. Several factors such as age, diabetes mellitus, hypertension, stenting of small coronary arteries, and ﬁnal total length of stents have been shown to be associated with an elevated risk of restenosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with CAD

Exclusion Criteria:

* PATIENTS WITHOUT OTHER HEALTH PROBLEMS

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study will include all patients with stable CAD who had previously undergone balloon angioplasty with stenting using drug-eluting stents that referred to the catheterization lab unit of Sohag University for recurrence of angina symptoms or positive cardiac tests. According to the results of the control angiography, the patients will be divided into two groups: patients with ISR confirmed by coronary angiography (angiographic restenosis of more than 50% of the target vessel) and patients without restenosis non ISR group. The patients with ISR were classified into subgroups by the terms of the restenosis development ( early before 12 months & late after 12 months).
Sampling Method: Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Angiotensin Converting Enzyme rs (1799752) gene polymorphism and Development of In-Stent Restenosis in Patients with Stable Coronary Artery Diseases | 2 months
  GENOTYPING of Converting Enzyme rs (1799752) gene in Development of In-Stent Restenosis in Patients with Stable Coronary Artery Diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne RA, Joner M, Kastrati A. Stent thrombosis and restenosis: what have we learned and where are we going? The Andreas Gruntzig Lecture ESC 2014. Eur Heart J. 2015 Dec 14;36(47):3320-31. doi: 10.1093/eurheartj/ehv511. Epub 2015 Sep 28. PMID 26417060
- [Background] Donisan T, Madanat L, Balanescu DV, Mertens A, Dixon S. Drug-Eluting Stent Restenosis: Modern Approach to a Classic Challenge. Curr Cardiol Rev. 2023;19(3):e030123212355. doi: 10.2174/1573403X19666230103154638. PMID 36597603
- [Background] Nakano M, Vorpahl M, Otsuka F, Taniwaki M, Yazdani SK, Finn AV, Ladich ER, Kolodgie FD, Virmani R. Ex vivo assessment of vascular response to coronary stents by optical frequency domain imaging. JACC Cardiovasc Imaging. 2012 Jan;5(1):71-82. doi: 10.1016/j.jcmg.2011.09.015. PMID 22239896
- [Background] Danilczyk U, Penninger JM. Angiotensin-converting enzyme II in the heart and the kidney. Circ Res. 2006 Mar 3;98(4):463-71. doi: 10.1161/01.RES.0000205761.22353.5f. PMID 16514079